CLINICAL TRIAL: NCT04822402
Title: COVID-19 Among Pregnant Women in Isolation and Women Hospitals in Assiut
Brief Title: COVID-19 Among Pregnant Women in Assiut
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Mohamed Mahmoud, Resident Doctor, Assiut University
Other Study IDs: COVID-19 among Pregnant Women
Record Dates: First submitted 2021-03-27; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Covid-19 in Pregnancy
Keywords: COVID-19; Pregnancy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is a new disease , little is known about COVID-19 during pregnancy and to the best of our knowledge no published studies in Assiut .

Aims of the Research :

1. To describe COVID-19 among pregnant women attending isolation and women hospitals in Assiut .
2. To identify comorbidities that may affect both maternal , fetal and neonatal outcomes .
3. To correlate between COVID-19 infection and maternal, fetal and neonatal outcomes .

DETAILED DESCRIPTION:
COVID-19 is the disease caused by a new corona virus on December 2019 in Wuhan, China . On February 2020, the International Committee of Taxonomy of Viruses recognized the etiology of this infection and named it "SARS-CoV-2". World Health Organization (WHO) named the disease COVID-19 , and declared it a pandemic on March 11th 2020 .

Pregnant women are at an increased risk for severe illness from COVID-19 compared to non-pregnant women . Additionally, pregnancy represents a vulnerable period, and this pandemic can negatively impact its outcomes . Therefore, pregnant women may be a group requiring special care in relation to the transmission of SARS-CoV-2 .

The modulations of the maternal immune system in pregnancy may have consequences for the clinical course of COVID-19 , for the treatment and prevention of COVID-19 in pregnancy . In addition to the systemic immunological changes, the reduction in total lung capacity and inability to clear secretions occurring during pregnancy can make pregnant more susceptible to severe respiratory infections .

There are higher levels of circulating coagulation and fibrinolytic factors during pregnancy which may be implicated in the pathogenesis of SARS-CoV-2 infection.

COVID-19 disease has a similar spectrum of symptoms in pregnant woman as in non-pregnant woman . Although most of the symptoms are less frequent during pregnancy but pregnant women are more likely to need admission to an ICU and require invasive ventilation .

Pre-existing maternal comorbidities such as increased maternal age, high body mass index, chronic hypertension and pre-existing diabetes are risk factors for the severity of infection.

The overall data from cohort studies by Allotey et al. , showed 73 deaths (0.63%) in COVID-19 positive pregnant women. The severe form of COVID-19 manifested in 13% of pregnant women, admission to an intensive care unit was required for 4% , 3% required invasive ventilation and 0.4% required extracorporeal membrane oxygenation .

Hsu et al. study on COVID-19 symptom progression during pregnancy compared to non pregnant women showed that 8.3% of the COVID-19 pregnant women had severe disease of whom 86% progressed to a critical stage and were admitted to the ICU , another study by Blitz et al. showed no significant difference between the rates of ICU admission in hospitalized COVID-19 pregnant and non-pregnant COVID-19 positive patients .

Vertical transmission happens if an infected pregnant woman transmits the infection to her fetus / infant during the fetal , intra-partum or post-partum period . Kotlyar et al. in their systematic review and meta-analysis showed a pooled proportion of 3.2% for vertical transmission of COVID-19 infection .

Other studies as Penfield et al. have shown a linkage of vertical transmission with maternal disease severity .

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with confirmed COVID-19 in Isolation hospitals in Assiut recorded and diagnosed by PCR swab from 1/3/2020 until the end of October 2021.

Exclusion Criteria:

* Pregnant women who are probably or suspected to be infected with COVID-19.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Descriptive cross-sectional study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Understanding of the epidemiology of COVID-19 in pregnancy . | baseline
  The understanding of the epidemiology of COVID-19 in pregnancy will provide critical data about the course of the disease in pregnant women and their infants .

SECONDARY OUTCOMES:
Developing a recommendations . | baseline
  Developing a recommendations relating to antenatal , intrapartum and postpartum care of women in order to help improvement the maternal and neonatal outcomes.

REFERENCES:
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Background] Sanchez-Sanchez E, Ramirez-Vargas G, Avellaneda-Lopez Y, Orellana-Pecino JI, Garcia-Marin E, Diaz-Jimenez J. Eating Habits and Physical Activity of the Spanish Population during the COVID-19 Pandemic Period. Nutrients. 2020 Sep 15;12(9):2826. doi: 10.3390/nu12092826. PMID 32942695
- [Background] Caparros-Gonzalez RA. [Maternal and neonatal consequences of coronavirus COVID-19 infection during pregnancy: a scoping review]. Rev Esp Salud Publica. 2020 Apr 17;94:e202004033. Spanish. PMID 32382001
- [Background] Silasi M, Cardenas I, Kwon JY, Racicot K, Aldo P, Mor G. Viral infections during pregnancy. Am J Reprod Immunol. 2015 Mar;73(3):199-213. doi: 10.1111/aji.12355. Epub 2015 Jan 13. PMID 25582523
- [Background] Goodnight WH, Soper DE. Pneumonia in pregnancy. Crit Care Med. 2005 Oct;33(10 Suppl):S390-7. doi: 10.1097/01.ccm.0000182483.24836.66. PMID 16215363
- [Background] Ji HL, Zhao R, Matalon S, Matthay MA. Elevated Plasmin(ogen) as a Common Risk Factor for COVID-19 Susceptibility. Physiol Rev. 2020 Jul 1;100(3):1065-1075. doi: 10.1152/physrev.00013.2020. Epub 2020 Mar 27. PMID 32216698
- [Background] Allotey J, Stallings E, Bonet M, Yap M, Chatterjee S, Kew T, Debenham L, Llavall AC, Dixit A, Zhou D, Balaji R, Lee SI, Qiu X, Yuan M, Coomar D, Sheikh J, Lawson H, Ansari K, van Wely M, van Leeuwen E, Kostova E, Kunst H, Khalil A, Tiberi S, Brizuela V, Broutet N, Kara E, Kim CR, Thorson A, Oladapo OT, Mofenson L, Zamora J, Thangaratinam S; for PregCOV-19 Living Systematic Review Consortium. Clinical manifestations, risk factors, and maternal and perinatal outcomes of coronavirus disease 2019 in pregnancy: living systematic review and meta-analysis. BMJ. 2020 Sep 1;370:m3320. doi: 10.1136/bmj.m3320. PMID 32873575
- [Background] Hsu AL, Guan M, Johannesen E, Stephens AJ, Khaleel N, Kagan N, Tuhlei BC, Wan XF. Placental SARS-CoV-2 in a pregnant woman with mild COVID-19 disease. J Med Virol. 2021 Feb;93(2):1038-1044. doi: 10.1002/jmv.26386. Epub 2020 Nov 10. PMID 32749712
- [Background] Blitz MJ, Grunebaum A, Tekbali A, Bornstein E, Rochelson B, Nimaroff M, Chervenak FA. Intensive care unit admissions for pregnant and nonpregnant women with coronavirus disease 2019. Am J Obstet Gynecol. 2020 Aug;223(2):290-291. doi: 10.1016/j.ajog.2020.05.004. Epub 2020 May 7. No abstract available. PMID 32387323
- [Background] Kotlyar AM, Grechukhina O, Chen A, Popkhadze S, Grimshaw A, Tal O, Taylor HS, Tal R. Vertical transmission of coronavirus disease 2019: a systematic review and meta-analysis. Am J Obstet Gynecol. 2021 Jan;224(1):35-53.e3. doi: 10.1016/j.ajog.2020.07.049. Epub 2020 Jul 31. PMID 32739398
- [Background] Penfield CA, Brubaker SG, Limaye MA, Lighter J, Ratner AJ, Thomas KM, Meyer JA, Roman AS. Detection of severe acute respiratory syndrome coronavirus 2 in placental and fetal membrane samples. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100133. doi: 10.1016/j.ajogmf.2020.100133. Epub 2020 May 8. No abstract available. PMID 32391518
- See also: World Health Organization Press Conference. The World Health Organization (WHO) Has Officially Named the Disease Caused by the Novel Coronavirus as COVID-19. [(accessed on 11 February 2020)] — http://www.who.int/emergencies/diseases/novel-coronavirus-2019